CLINICAL TRIAL: NCT06499090
Title: The Effect of Peri-operative Mirtazapine on Acute and Chronic Post Mastectomy Pain (Prospective Randomized Controlled Study)
Brief Title: Mirtazapine for Acute and Chronic Post Mastectomy Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Rabiee Ali, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: mirtazapine for post mastectoy
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mirtazapine group (Active Comparator): patients will receive orally the night before surgery the study medication and daily up to two weeks after: Mirtazapine group: Mirtazapine 30 mg tablet
  Interventions: Drug: Mirtazapine 30 MG
- placebo group (Placebo Comparator): patients will receive orally the night before surgery the study medication and daily up to two weeks after:
  placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine 30 MG — patients will receive orally the night before surgery the study medication and daily up to two weeks after Mirtazapine 30 mg tablet
  Arms: Mirtazapine group
Drug: Placebo — patients will receive orally the night before surgery the study medication and daily up to two weeks after placebo tablet
  Arms: placebo group

SUMMARY:
Our aim in this study will be to investigate the effect of mirtazapine on acute post-mastectomy pain manifested by total morphine consumption in first 24 hours and VAS score at rest and movement (primary outcomes). chronic neuropathic pain using LANSS Pain Scale (Leeds Assessment of Neuropathic Signs and Symptoms) and to evaluate the quality of recovery using the quality of recovery-40scoring system(QoR-40) (secondary outcomes) following modified radical mastectomy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

female patients aged 20-70 years scheduled for modified radical mastectomy with axillary dissection for breast carcinoma

Exclusion Criteria:

* known allergy to the study drugs significant organ dysfunction drug or alcohol abuse epilepsy patients with chronic pain or regularly receiving analgesics any psychiatric illness that would interfere with the perception and the assessment of pain

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 62 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
The cumulative postoperative 24 h morphine consumption | 24 hours

SECONDARY OUTCOMES:
The visual analogue score of pain intensity | 24 hours
  VAS score of pain intensity at rest and arm movement (abduction of the arm of the operated side up to 90°) measured at (0, 2,4,8,12,16 and 24h) postoperatively.
The quality of recovery-40 questionnaire | 24 hours
  1 means very poor recover and 40 very good recovery
Assessment of sedation level | 24 hours
  Assessment of sedation level by the Modiﬁed Ramsay Sedation score
Assessment of chronic pain | 6 months
  Assessment of chronic pain will be done after the first, third and Sixth month post-operatively by LANSS to evaluate chronic pain in the Pain Clinic.
Depression score | 6 months
  Depression score by the Patient Health Questionnaire(PHQ9)

CONTACTS AND LOCATIONS:
Locations (1):
- south Egypt Cancer Institute Assiut University, Asyut, Egypt

REFERENCES:
- See also: combination of mirtazapine and milnacipran augments the extracellular levels of monoamines in the rat brain. — https://pubmed.ncbi.nlm.nih.gov/22342987/